CLINICAL TRIAL: NCT02846155
Title: Gastric Preparation of Magnetic-controlled Capsule Endoscopy: A Prospective, Single Blinded and Randomized Controlled Trial
Brief Title: Gastric Preparation of Magnetic-controlled Capsule Endoscopy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, M.D., Associate Professor, Associate Chief Physician, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 20160410A
Record Dates: First submitted 2016-07-21; First posted 2016-07-27 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Stomach Diseases
Keywords: preparation; capsule endoscopy
MeSH Terms: conditions — Stomach Diseases | interventions — Simethicone; Pronase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- clear water group (Placebo Comparator): the patients only drink 1000ml clear water before checking
  Interventions: Other: clear water
- simethicone group (Experimental): the patients drink 950ml clear water and 15ml simethicone before checking
  Interventions: Drug: simethicone
- simethicone combined with pronase group (Experimental): the patients drink 900ml clear water and 15ml simethicone and 20，000iu pronase before checking
  Interventions: Drug: simethicone combined with pronase

INTERVENTIONS:
Other: clear water — the patients just drink common clear water before Magnetic-controlled Capsule Endoscopy examination
  Arms: clear water group
Drug: simethicone — the patients drink clear water and simethicone (Espumisan; Berlin-Chemie, Germany, containing 40 mg simethicone in 1 mL emulsion) before Magnetic-controlled Capsule Endoscopy examination
  Arms: simethicone group
Drug: simethicone combined with pronase — the patients drink simethicone (Espumisan; Berlin-Chemie, Germany, containing 40 mg simethicone in 1 mL emulsion)，pronase granules（Deyou；Beijing Tide Pharmaceutical Co，China,containing 20,000iu pronase），and clear water before Magnetic-controlled Capsule Endoscopy examination
  Arms: simethicone combined with pronase group

SUMMARY:
By using three different Gastric Preparation of Magnetic-controlled Capsule Endoscopy, the investigators hope to find out the optimal gastric preparation plan.

DETAILED DESCRIPTION:
It is a prospective, single-blind, randomized controlled trial. Patients who were conducted by Magnetic-controlled Capsule Endoscopy at Changhai Hospital will be randomly allocated into three different Gastric Preparation group before the procedure. It include clear water group which patient only drink 1000ml clear water before checking; simethicone group which patient drink 950ml clear water and 15ml simethicone before checking; simethicone combined with pronase group which patient drink 900ml lear water and 15ml simethicone and 20，000iu pronase before checking. The result were got from a relevant professional physician's blinded independent image-reading.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 16-75 years, who were scheduled to undergo a Magnetic-controlled Capsule Endoscopy, were eligible for this study.

Exclusion Criteria:

* Dysphagia or symptoms of gastric outlet obstruction, suspected or known intestinal stenosis, overt gastrointestinal bleeding, history of upper gastrointestinal surgery or abdominal surgery altering gastrointestinal anatomy, or postabdominal radiation;
* Congestive heart failure, renal insufficiency, under therapeutic anticoagulation, in poor general condition (American Society of Anesthesiologists class III/IV), claustrophobia, metallic parts, a pacemaker or other implanted electromedical devices, artificial heart valves;
* Pregnancy or suspected pregnancy;
* Exclusion criteria for standard magnetic resonance imaging (MRI) examination such as the presence of surgical metallic devices, even though its low magnetic field would technically not interfere with such devices;
* Currently participating in another clinical study.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
the level of gastric cleansing | 4 month
  Two investigators who did not know which kind of gastric preparation of the patient scored the level of gastric cleansing 0f 120 participants according to a four-point grading scale: poor, fair, good, and excellent，which was pointed 3,2,1，and 0.The investigators should evaluate the gastric cleansing of six anatomical landmarks (cardia, fundus, body, angulus, antrum and pylorus).A poor level of cleansing indicated the mucosa was obscured largely by a lot of air bubbles and grume,fair indicated that a portion of the mucosa was obscured by air bubbles and grume that was enough to prevent a reliable visualization of polyps, good indicated that a small amount of air bubbles and grume，and excellent indicated that the fluid was clear and the image was either free or had only small bits of air bubbles and grume.

SECONDARY OUTCOMES:
Transit time | 4 month
  include gastric transit time，smal bowel transit time
Diagnostic yield of Magnetic-controlled Capsule Endoscopy | 4 month
  The gastric focal lesion was defined as any of the positive findings including polyp, ulcers, submucosal tumor (SMT) and others (i.e. xanthoma, diverticulum, etc.). Erosion, gastritis and gastric atrophy were defined as negative findings, because they are diffuse lesions which can be easily diagnosed by Magnetic-controlled Capsule Endoscopy.
Tolerability of participants | 4 month
  The endoscopist scored the tolerability of participants according to a three-point grading scale: poor, fair, and excellent，which was pointed 2,1，and 0.A poor tolerability of participants indicated patients with perforated severe abdominal pain,nausea, vomiting，etc.fair indicated patients with perforated little abdominal pain,nausea, vomiting.and excellent indicated that patients with no obvious discomfort.
the visibility of gastric | 4 month
  Two investigators scored the level of gastric visibility 0f 120 participants according to a four-point grading scale: poor, fair, good, and excellent，which was pointed 3,2,1,and 0.The investigators should evaluate the visibility of gastric of six anatomical landmarks (cardia, fundus, body, angulus, antrum and pylorus).A poor level of cleansing indicated the less than 50% of mucosa could be seen,fair indicated that 50%-75% of the mucosa could be seen, good indicated that more than 75% of the mucosa could be seen，and excellent indicated the whole mucosa could be seen.
the time of gastric examination | 4 month
  the time indicated since the first gastric mucosal image was observed to the endoscopist completed the whole gastric examination。
the added amount of water of the whole process during gastric examination | 4 month

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided